CLINICAL TRIAL: NCT02010645
Title: Phase II Study of Eltrombopag in Combination With Decitabine in Subjects With Advanced Myelodysplastic Syndrome
Brief Title: Eltrombopag With Decitabine in Advanced Myelodysplastic Syndrome (MDS)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: PI Request
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2013-0590; NCI-2014-01276 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2013-12-05; First posted 2013-12-13 (Estimated); Results first posted 2020-01-02 (Actual); Last update posted 2020-01-02 (Actual); Status verified 2019-12

CONDITIONS: Leukemia
Keywords: Leukemia; Advanced Myelodysplastic Syndrome; MDS; Intermediate-2 Myelodysplastic Syndrome; High-Risk Myelodysplastic Syndrome; Chronic myelomonocytic leukemia; CMML; Eltrombopag; Promacta; Decitabine; Dacogen
MeSH Terms: conditions — Leukemia; Leukemia, Myelomonocytic, Chronic | interventions — eltrombopag; Decitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Eltrombopag + Decitabine (Experimental): Starting dose of Eltrombopag is 100 mg by mouth daily for each 28 day cycle. East Asians will start at 50 mg by mouth daily for each 28 day cycle.
  Starting dose of Decitabine is 20 mg/m2 by vein on Days 1-5 for each 28 day cycle.
  Interventions: Drug: Eltrombopag; Drug: Decitabine

INTERVENTIONS:
Drug: Eltrombopag — Starting dose of Eltrombopag is 100 mg by mouth daily for each 28 day cycle. East Asians will start at 50 mg by mouth daily for each 28 day cycle.
  Other Names: Promacta
Drug: Decitabine — Starting dose of Decitabine is 20 mg/m2 by vein on Days 1-5 for each 28 day cycle.
  Other Names: Dacogen

SUMMARY:
The goal of this clinical research study is to learn if eltrombopag given in combination with decitabine can help to control advanced MDS. The safety of this study drug combination will also be studied.

DETAILED DESCRIPTION:
Study Drug Administration:

Each cycle is 28 days.

If you are found to be eligible to take part in this study, you will receive decitabine by vein over 1 hour on Days 1-5 of each cycle.

You will also take eltrombopag capsules by mouth 1 time every day of each cycle. You should take it on an empty stomach (1 hour before a meal or 2 hours after a meal) with 8 ounces (1 cup) of water.

Do not eat calcium-rich foods (such as dairy products and juices with added calcium), or take other drugs (such as antacids) or supplements containing iron, calcium, aluminum, magnesium, selenium, and/or zinc for 4 hours before or 4 hours after taking eltrombopag.

If a dose of eltrombopag is vomited, you should not make it up or re-take it on the same day. If the morning dose is missed, it may be taken up until 5:00 PM on the same day.

Study Visits:

On Day 1 of each cycle:

* You will have a physical exam.
* Blood (about 2-3 teaspoons) will be drawn for routine tests.

On Days 8, 15, and 22 of Cycle 1 only, blood (about 2-3 teaspoons) will be drawn for routine tests.

If the doctor thinks it is needed, on Day 1 of Cycles 2-4, then every 3 cycles (Cycles 7, 10, 13, and so on), you will also have a bone marrow aspirate/biopsy to check the status of the disease and for cytogenetic testing.

If the doctor thinks it is needed, once each week blood (about 2-3 teaspoons) will be drawn for routine tests.

End-of-Treatment Visit:

Within 5 days of your last dose of study drug, you will come to the clinic for an end-of-treatment visit. The following procedures will be performed:

* You will have a physical exam.
* Blood (about 2-3 teaspoons) will be drawn for routine tests.
* You will have a bone marrow aspirate/biopsy to check the status of the disease and for cytogenetic testing.

Length of Study:

You may continue taking the study drugs for as long as the doctor thinks it is in your best interest. You will no longer be able to take the study drugs if the disease gets worse, if intolerable side effects occur, or if you are unable to follow study directions.

Your participation on the study will be over after the follow-up visits.

Follow-up Visit:

About 28 days after your last dose of study drugs, you will come to the clinic for a follow-up visit. The following procedures will be performed:

* You will have a physical exam.
* Blood (about 2-3 teaspoons) will be drawn for routine tests.

This is an investigational study. Eltrombopag is FDA approved and commercially available for the treatment of low platelet counts in patients with idiopathic thrombocytopenic purpura (ITP -- a severe bleeding disease). Decitabine is FDA approved for the treatment of MDS and is commercially available. The combination of eltrombopag and decitabine to treat MDS is investigational.

Up to 50 patients will take part in this study. All will be enrolled at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Signed, informed consent must be obtained prior to any study specific procedures.
2. Subjects with a histologically confirmed diagnosis of MDS by FAB criteria, including both MDS and RAEB-T (AML with 20-30% blasts and multilineage dysplasia) and chronic myelomonocytic leukemia (CMML) with at least 10% bone marrow blasts by World Health Organization (WHO) classification are eligible.
3. Advanced MDS by virtue of intermediate-2 or high-risk MDS by IPSS score, or high or very-high risk by IPSS-R.
4. Platelet count </= 100 x 10^9/L at baseline
5. Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 2
6. Adequate liver function, as evidenced by a serum bilirubin </= 2x the ULN (except for patients with a confirmed diagnosis of Gilbert's Disease) and an ALT or AST </= 3x the laboratory ULN.
7. Serum creatinine </= 2.5x upper limit of normal
8. Subjects must be >/= 18 years of age at the time of informed consent
9. Subject is practicing an acceptable method of contraception (documented in chart). Female subjects (or female partners of male subject) must either be of non-childbearing potential (hysterectomy, bilateral oophorectomy, bilateral tubal ligation or post-menopausal > 1 year), or of childbearing potential and use one of the following highly effective methods of contraception (i.e. Pearl index < 1.0%) from 2 weeks prior to administration of study medication, throughout the study, and 28 days after completion or premature discontinuation from the study: - Complete abstinence from intercourse; - Intrauterine device (IUD); - Two forms of barrier contraception (diaphragm plus spermicide, and for males condom plus spermicide); - Male partner is sterile prior to entry into the study and is the only partner of the female; - Systemic contraceptives (combined or progesterone only).

Exclusion Criteria:

1. Subjects with any prior exposure to a thrombopoietin-receptor agonist
2. Prior hypomethylating agent treatment for MDS
3. Any prior or co-existing medical condition that in the investigator's judgment will substantially increase the risk associated with the subject's participation in the study
4. Psychiatric disorders or altered mental status precluding understanding of the informed consent process and/or completion of the necessary study procedures
5. Active uncontrolled serious infection or sepsis at study enrollment
6. Clinically significant gastrointestinal disorders that may interfere with absorption of drug.
7. History of arterial thrombosis (i.e. stroke) in the past year
8. History of venous thrombosis currently requiring anti-coagulation therapy
9. Unstable angina, congestive heart failure (New York Heart Association (NYHA) > Class II), uncontrolled hypertension (diastolic blood pressure > 100mmHg), or recent (within 1 year) myocardial infarction
10. Subjects with a QTc > 480 msec (QTc > 510 msec for subjects with Bundle Branch Block) at baseline
11. Pregnant or breast-feeding
12. Subjects with known history of human immunodeficiency virus (HIV) or active infection with hepatitis C virus (HCV) or hepatitis B virus (HBV), because eltrombopag is hepatically cleared, and underlying hepatic impairment may lead to an increased risk of hepatotoxicity. Eltrombopag has not been evaluated with combination antiretroviral regimens.
13. Subjects with liver cirrhosis (as determined by the investigator)
14. Subjects with hypersensitivity to study drugs or their excipients.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2014-03 (Actual); Primary Completion 2019-01-02 (Actual); Study Completion 2019-01-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Courtney DiNardo, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment period: March 2014 to February 2015
Groups:
- Eltrombopag + Decitabine: Starting dose of Eltrombopag is 100 mg by mouth daily for each 28 day cycle. East Asians will start at 50 mg by mouth daily for each 28 day cycle.
  Starting dose of Decitabine is 20 mg/m2 by vein on Days 1-5 for each 28 day cycle.
  Eltrombopag: Starting dose of Eltrombopag is 100 mg by mouth daily for each 28 day cycle. East Asians will start at 50 mg by mouth daily for each 28 day cycle.
  Decitabine: Starting dose of Decitabine is 20 mg/m2 by vein on Days 1-5 for each 28 day cycle.
Period: Overall Study
Arm/Group | Eltrombopag + Decitabine
Started | 6
Completed | 6
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Eltrombopag + Decitabine
Number analyzed (Participants) | 6
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 2
  >=65 years | 4
Age, Continuous [Median (Full Range); unit: years] | 75 [56 to 78]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 6
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 6

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate (ORR)
Description: The primary endpoint is the overall response rate (ORR) based on the IWG-2006 criteria, which includes complete remission (CR), partial remission (PR), and hematologic improvement (HI).
Time Frame: 28 days
Population: One participant was not evaluable for response.
Measure: Count of Participants; unit: Participants
Arm/Group | Eltrombopag + Decitabine
Number analyzed (Participants) | 5
Participants | 1

ADVERSE EVENTS:
Time Frame: 3 years and 9 months
Arm/Group | Eltrombopag + Decitabine
All-Cause Mortality (participants affected / at risk) | 1/6
Serious Adverse Events (participants affected / at risk) | 4/6
Other Adverse Events (participants affected / at risk) | 5/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Eltrombopag + Decitabine (N=6)
Lung Infection (Infections and infestations) | 1 (1)
Neutropenic Fever (Infections and infestations) | 2 (2)
Flank Pain (General disorders) | 1 (1)
Fall (General disorders) | 1 (1)
Hyperbilirubinemia (Metabolism and nutrition disorders) | 1 (1)
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Retroperitoneal Hemorrhage (Gastrointestinal disorders) | 1 (1)
Cardiac Arrest (Cardiac disorders) | 1 (1)
Small Intestinal Obstruction (Gastrointestinal disorders) | 1 (1)
Portal Vein Thrombosis (Hepatobiliary disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Eltrombopag + Decitabine (N=6)
Back Pain (General disorders) | 1 (1)
Blurred Vision (Eye disorders) | 2 (3)
Colitis (Gastrointestinal disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (3)
Dizziness (Nervous system disorders) | 2 (2)
Fatigue (General disorders) | 2 (3)
Oral Mucositis (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 3 (3)
Neutropenia (Investigations) | 1 (1)
Palpitations (Cardiac disorders) | 1 (1)
Paresthesia (Nervous system disorders) | 1 (1)
Erythematous Rash (Skin and subcutaneous tissue disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2013-12-13): https://cdn.clinicaltrials.gov/large-docs/45/NCT02010645/Prot_SAP_000.pdf